CLINICAL TRIAL: NCT01441011
Title: Group Phone-Based Weight Control for Rural Breast Cancer Survivors
Brief Title: Rural Women Connecting for Better Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12633; 1R01CA155014-01A1 (NIH)
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer; Obesity
Keywords: weight loss; breast cancer; obesity; overweight; rural women; community based; Secondary Prevention
MeSH Terms: conditions — Breast Neoplasms; Obesity; Weight Loss; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group (GRP) phone counseling (Experimental): The group phone counseling includes 26 bi-weekly phone sessions from 6 to 18 months and focuses on group problem-solving. Women continue in the same group as in weight loss intervention phase.
  Interventions: Behavioral: Group phone counseling
- Mail-based Comparison Condition (Active Comparator): Participants in this group will receive a newsletter by mail every other week for 12 months starting after the initial 6 month weight loss period. The newsletters will provide problem-solving tips and will review nutrition and physical activity information.
  Interventions: Behavioral: Newsletter

INTERVENTIONS:
Behavioral: Group phone counseling — Bi-weekly phone counseling sessions from 6 - 18 months
  Arms: Group (GRP) phone counseling
Behavioral: Newsletter — Bi-weekly newsletter mailings from 6 - 18 months
  Arms: Mail-based Comparison Condition

SUMMARY:
Women who are obese at breast cancer diagnosis have a 1.5 to 2.5 increased risk of recurrence and death compared to their normal weight counterparts. Moreover, weight gain and decreased physical activity are common after diagnosis and also increase the likelihood of breast cancer recurrence and death. Rural women suffer from health disparities in breast cancer diagnosis and treatment. Women of the most rural counties also have the highest prevalence of obesity compared to urban women. To address these disparities, the overarching objective of this proposal is to develop a clinically effective and cost efficient strategy for delivering a weight control intervention to rural breast cancer survivors. Group phone-based treatment via conference call is a novel treatment delivery approach that the investigators have shown to be effective for initial weight loss among rural breast cancer survivors and more effective than the standard individual phone-based approach among rural women. This innovative method of providing group treatment addresses access barriers in rural areas and may be especially ideal for rural breast cancer survivors because it provides social support in conjunction with a level of anonymity. However, the impact of group phone counseling during extended care for weight loss maintenance beyond 6 months remains unknown. Weight loss maintenance is the more challenging phase of treatment when weight regain is common, and this regain presents a potential risk for breast cancer recurrence. This randomized controlled trial will evaluate the effects of group phone-based treatment for weight loss maintenance among rural breast cancer survivors, compared to an established mail-based education comparison condition, subsequent to a 6 month group phone-based weight loss phase for both conditions. In addition to the intervention impact on weight loss maintenance, the study will provide estimates of incremental cost-effectiveness per kg loss between the two conditions and the impact on secondary outcomes including quality of life, breast cancer risk biomarkers, dietary intake, and physical activity.

DETAILED DESCRIPTION:
Phase 1 - Weight Loss (0-6 months)

* Weekly group phone counseling sessions for all participants (12-14 women per group) via conference call for 26 consecutive weeks
* Low-calorie, low-fat diet recommended, including 2 pre-packaged entrees, five one-cup servings of fruits and vegetables and meal replacement shakes (provided free of charge)
* Physical activity program program recommended, beginning with 15 minutes per day, 3 days a week, working toward a goal of 225 minutes a week
* Experienced group counselor facilitates all sessions

Phase 2 - Weight Loss Maintenance (6-18 months)

* Participants randomized to either group phone counseling or mail-based comparison with no phone counseling
* Weight loss maintenance group condition includes 26 bi-weekly phone sessions, while mail-based comparison includes 26 bi-weekly newsletters in the mail
* Focus is on problem-solving

Phase 3 - Transition to Self-Reliance (18-24 months)

* Lasts from 18-24 months
* No sessions or newsletter mailings
* Participants are encouraged to continue to self-monitor throughout this period

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with a BMI 27-45 kg/m2
* Diagnosis of Stage 0-IIIc disease within the past 10 years (except Stage 0, treated with mastectomy only)
* Have completed all local and systemic therapy at least 3 months prior to entry
* Have clearance from their oncologist or current medical provider to participate in a weight control study
* Must be ≤ 75 years old
* Post-menopausal
* Participants must live in a rural area
* Have access to a phone
* Able to participate in the physical activity component of the intervention, i.e., be able to walk briskly unassisted and without serious medical risk
* Weight stable within ten pounds three months prior to entry

Exclusion Criteria:

* Women with insulin-dependent diabetes
* Ongoing participation in a formal weight loss program
* Ongoing use of pharmacotherapy for weight loss
* Ongoing use of medications that seriously affect weight and metabolism (e.g., steroids, phentermine)
* Positive screen for current substance abuse, major depression, or binge eating disorder
* Any cardiac or pulmonary disease preventing participation
* Treatment for any other cancers within the past year
* Previous bariatric surgery

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Weight loss maintenance | 6 - 18 months
  Examine the impact of group phone-based treatment on weight loss maintenance from 6 to 18 months, compared to a mail-based education COMPARISON condition, following a 6-month weight loss phase among obese rural breast cancer survivors.

SECONDARY OUTCOMES:
Quality of life | Baseline and 6, 12, 18, and 24 months
  Compare the effects of treatment conditions on aspects of quality of life important for breast cancer survivorship, including general physical, social, and emotional well-being, fatigue, arthralgia, lymphedema symptoms, menopausal symptoms, and depressive symptoms.
Breast cancer risk biomarkers | Baseline and 6 and 18 months
  Examine the association of weight change with changes in selected breast cancer risk biomarkers, including bioavailable estradiol, testosterone, and fasting insulin. Examine whether modulation of biomarkers is sustained during weight loss maintenance.
Cost effectiveness | 18 months
  Compare the incremental cost-effectiveness of weight loss maintenance (kg below baseline) between group and control conditions. Costs include fixed and variable provider costs (facility, time, phone charges, supplies) and fixed and variable participant costs (time, out-of-pocket expenses).

CONTACTS AND LOCATIONS:
Overall Officials: Christie Befort, Ph.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Fazzino TL, Fabian C, Befort CA. Change in Physical Activity During a Weight Management Intervention for Breast Cancer Survivors: Association with Weight Outcomes. Obesity (Silver Spring). 2017 Nov;25 Suppl 2(Suppl 2):S109-S115. doi: 10.1002/oby.22007. PMID 29086523
- [Derived] Fazzino TL, Fleming K, Befort C. Alcohol Intake Among Breast Cancer Survivors: Change in Alcohol Use During a Weight Management Intervention. JMIR Cancer. 2016 Nov 9;2(2):e15. doi: 10.2196/cancer.6295. PMID 28410181
- [Derived] Fazzino TL, Sporn NJ, Befort CA. A qualitative evaluation of a group phone-based weight loss intervention for rural breast cancer survivors: Themes and mechanisms of success. Support Care Cancer. 2016 Jul;24(7):3165-73. doi: 10.1007/s00520-016-3149-7. Epub 2016 Mar 2. PMID 26932848
- [Derived] Befort CA, Klemp JR, Fabian C, Perri MG, Sullivan DK, Schmitz KH, Diaz FJ, Shireman T. Protocol and recruitment results from a randomized controlled trial comparing group phone-based versus newsletter interventions for weight loss maintenance among rural breast cancer survivors. Contemp Clin Trials. 2014 Mar;37(2):261-71. doi: 10.1016/j.cct.2014.01.010. Epub 2014 Jan 31. PMID 24486636
- See also: National Cancer Institute: Cancer Survivorship Research — http://cancercontrol.cancer.gov/ocs/index.html